CLINICAL TRIAL: NCT01094314
Title: Impact of Culture Medium on Embryo Quality
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Gasthuisberg (Other)
Responsible Party: Thomas D'Hooghe, Prof, MD, PhD, University Hospital Gasthuisberg Leuven
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: ML4562
Record Dates: First submitted 2010-03-25; First posted 2010-03-26 (Estimated); Last update posted 2010-03-26 (Estimated); Status verified 2010-03

CONDITIONS: Embryo Development

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- sequential medium (Active Comparator)
  Interventions: Other: embryo culture medium
- single medium (Active Comparator)
  Interventions: Other: embryo culture medium

INTERVENTIONS:
Other: embryo culture medium — comparison between two types of embryo culture medium

SUMMARY:
The purpose of this study is to compare two culture media.

ELIGIBILITY:
Inclusion Criteria:

* Embryos of patients younger than 36 years old

Exclusion Criteria:

* Embryos of patients older than 36 years old

Ages: 1 Day to 3 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 790 (Estimated)
Dates: Start 2008-01; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
embryo quality: number and size of blastomeres, degree of fragmentation | day 1 -day 3

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Leuven, Catholic University Leuven, Leuven, Belgium

REFERENCES:
- [Derived] Paternot G, Debrock S, D'Hooghe TM, Spiessens C. Early embryo development in a sequential versus single medium: a randomized study. Reprod Biol Endocrinol. 2010 Jul 7;8:83. doi: 10.1186/1477-7827-8-83. PMID 20609226